CLINICAL TRIAL: NCT03774420
Title: Post-Operative Cognitive Dysfunction After Breast Surgery: Incidence and Relation With Common Intraoperative Neuromonitoring Data and Concentration of Propofol and Remifentanil Infused With Targeted Controlled Infusion (TCI )in Women With Laryngeal Mask Airway
Brief Title: Post Operative Cognitive Dysfunction After Breast Surgery
Status: Recruiting | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, Principal Investigator, University of Padova
Other Study IDs: MAST
Record Dates: First submitted 2018-11-15; First posted 2018-12-13 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Emergence Delirium; Post-Operative Cognitive Dysfunction
Keywords: Infusion pumps; Intraoperative brain monitoring
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim of this trial is to define if Post-Operative Cognitive Dysfunction, detected analyzing changes between pre-operative and post-operative Neurocognitive Test, and Postoperative Delirium, relate to concentration of effector's site concentration of propofol and remifentanil TCI and to the common intraoperative neuromonitoring values as well as to Pupillometry values (in particular Pupil Diameter, Pupil Latency, and Maximum Contraction Velcoity).

DETAILED DESCRIPTION:
Post-Operative Cognitive Dysfunction has not been yet investigated after general anaesthesia with Targeted-Controlled-Infusion (TCI) and Laryngeal-Mask-Airway (LMA), daily used in the investigator's Hospital to anesthetize women undergoing breast surgery. Aim of this trial is to define if neurocognitive tests (Montreal Cognitive Assessment, Trail Making Test A and B, Digit Span Test) before and after surgery, and CAM for Postoperative Delirium relate to concentrations at effector's site (Ce) of propofol and remifentanil TCI and the values of Bispectral Index and Entropy monitoring and Surgical Plethysmographic Index (SPI), as well as to Pupillometry values.

ELIGIBILITY:
Inclusion Criteria:

* General Anaesthesia delivered with Propofol and Remifentanil with Targeted Controlled Infusion
* Use of Laryngeal Mask airway

Exclusion Criteria:

* Neurological pathologies
* Haemodynamical instability during surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women subjected to breast surgery in general anaesthesia with Laryngeal-Mask-Airway (LMA) anesthetized with propofol and remifentanil delivered by Targeted-Controlled-Infusion (TCI) pumps. Women will be subjected to neurocognitive tests (GEMS, TMT A and B) the day before surgery and before hospital discharge. These test will be related to propofol and remifentanil concentrations at effector site during surgery and awakening, to BIS and Entropia values and to SPI and pupillometry values.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-Operative Cognitive Dysfunction in breast-surgery patients detected with Montreal Cognitive Assessment test | Patients will be subjected to Global Examination of Mental Test (GEMS) test one day before surgery and 1 day after surgery.
  Discover incidence of Post-Operative Cognitive decline analyzing changes in Post-Operative Cognitive Dysfunction changes between Pre-operative Global Examination of Mental Test (GEMS) test. Better neurocognitve outcome with higher scores)
Incidence of Post-Operative Cognitive Dysfunction in breast-surgery patients detected with Trail Making Test A and B | Patients will be subjected to Trail Making Test (TMT) A and B one day before surgery and 1day after surgery.
  Discover Post-Operative Cognitive Dysfunction analyzing changes between Pre-operative Trail Making Test A and B test score and post-operative Trail Making Test A and B test score. These tests will be evaluated in seconds required to be completed (better neurocognitive outcome with fewer seconds required)
Incidence of Post-Operative Delirium in breast-surgery patients | Patients will be subjected to Confusion Assessment Method (CAM) within 1 hour from awakening from anesthesia .
  Discover Post-Operative Delirium submitting patients Confusion Assessment Method (CAM-ICU) test. Worse neurocognitve outcome with higher scores (ranging from 0 to 4)
Incidence of Post-Operative Cognitive Dysfunction in breast-surgery patients | Patients will be subjected to Short Portable Mental Status Questionnaire one day before surgery and 1 day after surgery.
  Discover Post-Operative Cognitive Dysfunction analyzing changes between Pre-operative Short Portable Mental Status Questionnaire score and post-operative Short Portable Mental Status Questionnaire test score. Better neurocognitve outcome with higher scores (ranging 0 to 10)
Incidence of Post-Operative Cognitive Dysfunction in breast-surgery patients detected with MiniMental State Evaluation test | Patients will be subjected to Confusion Assessment Method (CAM) within 1 hour from awakening from anesthesia.
  Discover Post-Operative Cognitive Dysfunction analyzing changes between Pre-operative Mini Mental State Evaluation test and postoperative Mini Mental State Evaluation test score. Worse eurocongitive outcome with lower scores.
Incidence of Emergence Delirium in breast-surgery patients detected with 4AT test | Patients will be subjected to 4 AT test within 1 day from awakening from anesthesia .
  Discover Post-Operative Cognitive Dysfunction analyzing acute changes in postoperative congition function utilizing the 4AT test. Worse neurocognitve outcome with higher scores. Worse neurocognitve outcome with higher scores

CONTACTS AND LOCATIONS:
Overall Officials: Federico Linassi, MD, Principal Investigator — University of Padova
Locations (1):
- Treviso Regional Hospital, Treviso, TV, Italy